CLINICAL TRIAL: NCT01695473
Title: A Pharmacodynamic Study of Pre-prostatectomy BKM120 in Men With High-risk, Localized Prostate Cancer
Brief Title: Neoadjuvant BKM120 in High-risk Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Accrual
Sponsor: Won Kim (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Won Kim, Prinicipal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 115516; NCI-2013-01830 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2012-09-26; First posted 2012-09-28 (Estimated); Results first posted 2021-01-13 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: High Risk Prostate Cancer
Keywords: Prostate cancer; High-risk prostate cancer; Radical prostatectomy; BKM120
MeSH Terms: conditions — Prostatic Neoplasms | interventions — NVP-BKM120

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant BKM120 (Experimental): Two weeks after confirmatory biopsy, patients will begin taking 100 mg/day of BKM120. BKM120 will be given at this dose level orally once daily for 14 days prior to radical prostatectomy. Radical prostatectomy will be performed on the day of the last dose of BKM120 at day 14. No further drug will be administered after radical prostatectomy. For unforeseen delays in operating room (OR) scheduling, up to 7 additional days of BKM120 may be administered prior to surgery.
  Interventions: Drug: BKM120

INTERVENTIONS:
Drug: BKM120 — Two weeks after confirmatory biopsy, patients will begin taking 100 mg/day of BKM120. BKM120 will be given at this dose level orally once daily for 14 days prior to radical prostatectomy. Radical prostatectomy will be performed on the day of the last dose of BKM120 at day 14. No further drug will be administered after radical prostatectomy. For unforeseen delays in OR scheduling, up to 7 additional days of BKM120 may be administered prior to surgery.
  Other Names: Buparlisib

SUMMARY:
This is a phase II, study of BKM120 in patients with high-risk, localized prostate cancer. Eligible patients will be enrolled and scheduled to have an ultrasound-guided biopsy of the prostate to confirm high-risk disease and collect prostate tissue for analysis. Two weeks after the biopsy, patients will begin taking 100 mg/day of BKM120. BKM120 will be given at this dose level orally once daily for 14 days prior to radical prostatectomy at University of California, San Francisco. Radical prostatectomy will be performed on the day of the last dose of BKM120 at day 14. No further drug will be tken after the radical prostatectomy.

DETAILED DESCRIPTION:
This is a phase II, prospective, pharmacodynamic study of BKM120 in high-risk, localized prostate cancer. After informed consent and central pathology review of the core prostate biopsy, eligible patients will be enrolled and scheduled to have an ultrasound-guided biopsy of the prostate to confirm high-risk disease and collect tissue for molecular analysis. Two weeks after the biopsy, patients will begin taking 100 mg/day of BKM120. BKM120 will be given at this dose level orally once daily for 14 days prior to radical prostatectomy at University of California, San Francisco. Radical prostatectomy will be performed on the day of the last dose of BKM120 at day 14. No further drug will be administered after radical prostatectomy.

Up to 24 patients, or 21 evaluable patients, will be enrolled through the Department of Urology or Genitourinary Medical Oncology at the University of California, San Francisco for this pharmacodynamic study. Toxicity will be assessed during BKM120 administration, and will involve a clinic visit on Day 14 ± 2 (i.e. before surgery). Follow-up with safety evaluations will be at 90 ± 7 days post-operatively and involve a toxicity questionnaire, blood tests, and clinic visit. Toxicity will be monitored and reported using NCI Common Toxicity Criteria version 4.0 guidelines.

A patient symptom diary will be distributed to each patient at baseline for symptom self-recording and BKM120 dose self-administration. In addition, a patient identifier card (wallet-sized) will be distributed to each patient after informed consent and registration. This information will contain the patient's age, study name and number, investigator and study coordinator contact information, and expected adverse events that may be present as a result of BKM120 administration.

ELIGIBILITY:
INCLUSION CRITERIA

1. Histologically confirmed adenocarcinoma of the prostate
2. Candidate for radical prostatectomy
3. Prostate cancer with the following pathological characteristics:

   1. Gleason sum > 8 AND at least 2 discrete core biopsies containing a minimum of 20% cancer or,
   2. Gleason pattern 4 + 3 = 7 and greater than 50% of biopsies positive for prostate cancer
4. Age >= 18 years
5. Eastern Cooperative Oncology Group (ECOG) performance status > 2
6. Ability to take oral medications (capsule must be swallowed with liquid)
7. Adequate bone marrow function as shown by: Absolute Neutrophil Count (ANC) >= 1.5 x 109/liter, Platelets ≥ 100 x 109/L, Hemoglobin > 9 grams(g) /decilitre(dL)
8. Total calcium (corrected for serum albumin) within normal limits (biphosphonate use for malignant hypercalcemia control is not allowed)
9. Magnesium >= the lower limit of normal
10. Potassium within normal limits for the institution
11. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) within normal range
12. Serum bilirubin within normal range (or total bilirubin <= 3.0 x upper limit of normal (ULN) with direct bilirubin within normal range in patients with well documented Gilbert Syndrome)
13. Serum creatinine <= 1.5 x upper limit of normal (ULN) or 24-hour clearance >= 50 milliliter per min (mL/min)
14. Serum amylase <= ULN
15. Serum lipase <= ULN
16. Fasting plasma glucose <= 120 mg/dL (6.7 mmol/L)
17. International Normalized Ratio (INR) <= 2
18. Men of reproductive potential and their female partners must use highly effective contraception during treatment, for 5 half-lives (8 days) after stopping treatment and for additional 12 weeks (3 months in total after study drug discontinuation) and should not father a child in this period The highly effective contraception is defined as either:

    1. True abstinence: When this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
    2. Sterilization: Female partners have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
    3. Male participant sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate).
    4. Use of a combination of any two of the following (a+b):
    5. Female partner with prior placement of an intrauterine device (IUD) or intrauterine system (IUS)
    6. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository • Oral contraception use by female partners, injected or implanted hormonal methods are not allowed as BKM120 potentially decreases the effectiveness of hormonal contraceptives.

       * Fertile males, defined as all males physiologically capable of conceiving offspring must use condom during treatment, for 5 half-lives (8 days) after stopping treatment and for additional 12 weeks (3 months in total after study drug discontinuation) and should not father a child in this period.
19. Ability to understand and the willingness to sign a written informed consent document

EXCLUSION CRITERIA

1. Prior treatment with a phosphatidylinositol 3-kinase (PI3K) inhibitor
2. Known hypersensitivity to BKM120 or to its excipients
3. History of another malignancy within 3 years, except cured basal cell carcinoma of the skin
4. Hormonal therapy with Gonadotropin-releasing hormone (GnRH) agonists, GnRH antagonists or high dose bicalutamide within 1 month of enrollment unless serum testosterone is within normal limits.
5. Following mood disorders as judged by the investigator and/or symptom management service co-investigator, or as a result of patient's mood assessment questionnaire:

   • Medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (immediate risk of doing harm to others)

   • Current >= NCI Common Terminology Criteria for Adverse Events (CTCAE) grade 3 anxiety

   • Meets the cut-off score of >= 10 in the Patient Health Questionnaire (PHQ-9) or a cut-off of >= 15 in the Generalized Anxiety Disorder (GAD-7) mood scale, respectively, or selects a positive response of "1, 2, or 3" to question number 9 regarding potential for suicidal thoughts in the PHQ-9 (independent of the total score of the PHQ-9) will be excluded from the study
6. Current diarrhea >= CTCAE grade 2
7. Active cardiac disease including any of the following:

   • History of left ventricular ejection fraction (LVEF) < 50% as determined by Multiple Grated acquisition (MUGA) scan or echocardiogram (ECHO)

   • QTc > 450 msec on screening electrocardiogram (ECG (using the QTcF formula)
   * Angina pectoris that requires the use of anti-anginal medication
   * History of ventricular arrhythmias except for benign premature ventricular contractions
   * Supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication
   * Conduction abnormality requiring a pacemaker
   * Valvular disease with documented compromise in cardiac function
   * Symptomatic pericarditis
8. History of cardiac dysfunction including any of the following:

   * Myocardial infarction within the last 6 months, documented by persistent elevated cardiac enzymes or persistent regional wall abnormalities on assessment of LVEF function
   * History of documented congestive heart failure (New York Heart Association functional classification III-IV)
   * Documented cardiomyopathy
9. Poorly controlled diabetes mellitus or active, steroid-induced diabetes mellitus
10. Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g., active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with the protocol
11. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of BKM120 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection). Patients with unresolved diarrhea will be excluded as previously indicated
12. Treatment with any hematopoietic colony-stimulating growth factors (G-CSF or GM-CSF) <= 2 weeks prior to starting study drug. Erythropoietin or darbepoetin therapy, if initiated at least 2 weeks prior to enrollment, may be continued
13. Current treatment with medication with a known risk to prolong the QT interval or inducing Torsades de Pointes and the treatment cannot either be discontinued or switched to a different medication prior to starting study drug. Please refer to section 10.2 for a list of prohibited QT prolonging drugs with risk of Torsades de Pointes.
14. Current, chronic treatment with steroids or another immunosuppressive agent

    • Note: Topical applications (e.g. rash), inhaled sprays (e.g. obstructive airways diseases), eye drops or local injections (e.g. intr-articular) are allowed. If a patient stops corticosteroids prior to study participation, a 2-week washout is required.
15. Taking herbal medications and certain fruits and juices within 7 days prior to starting study drug. Herbal medications include, but are not limited to St. John's wort, Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng. Fruits and juice include the Cytochrome P450 3A (CYP3A) inhibitors: Seville oranges, grapefruit, and pomelos.
16. Current treatment with drugs known to be moderate and strong inhibitors or inducers of isoenzyme CYP3A, and the treatment cannot be discontinued or switched to a different medication prior to starting study drug. Please refer to Section 10.2 for a list of prohibited inhibitors and inducers of CYP3A (Please note that co-treatment with weak inhibitors of CYP3A is allowed)
17. Chemotherapy or targeted anticancer therapy ≤ 4 weeks (6 weeks for nitrosourea, antibodies or mitomycin-C) prior to starting study drug
18. Any continuous or intermittent small molecule therapeutics (excluding monoclonal antibodies) <= 5 effective half lives prior to starting study drug or patients who have not recovered from side effects of such therapy 19 Major surgery <= 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy

20. Current treatment with warfarin sodium or any other coumadin-derivative anticoagulant 21. Known diagnosis of human immunodeficiency virus (HIV) infection. Testing is not required for participation.

22. Unable or unwilling to abide by the study protocol or cooperate fully with the investigator

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-04-23 (Actual); Primary Completion 2015-02-05 (Actual); Study Completion 2015-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Won Kim, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Neoadjuvant BKM120: Two weeks after confirmatory biopsy, patients will begin taking 100 mg/day of BKM120. BKM120 will be given at this dose level orally once daily for 14 days prior to radical prostatectomy. Radical prostatectomy will be performed on the day of the last dose of BKM120 at day 14. No further drug will be administered after radical prostatectomy. For unforeseen delays in OR scheduling, up to 7 additional days of BKM120 may be administered prior to surgery.
Period: Overall Study
Arm/Group | Neoadjuvant BKM120
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Neoadjuvant BKM120
Number analyzed (Participants) | 11
Age, Continuous [Mean (Full Range); unit: Years] | 61 [53 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 11
Pre-treatment Prostate-specific antigen (PSA) [Median (Full Range); unit: nanograms per mililiter (ng/mL)] | 21.7 [5.7 to 146.3]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Decrease in Phosphorylated S6 Immunohistochemistry (ICH) From Baseline
Description: Percentage of men with downstream target inhibition of PI3K in prostate tumor tissue as measured by phosphorylated S6 immunohistochemistry (ICH) when treated with 100 mg/day of BKM120 using paired tumor biopsies from before and after drug administration and defined as ≥ 60% decrease in phosphorylated S6 (pS6) from baseline by Immunohistochemistry (IHC).
Time Frame: Up to 3 months
Population: One patient did not have pretreatment tissue evaluable for IHC
Measure: Number; unit: percentage of participants
Arm/Group | Neoadjuvant BKM120
Number analyzed (Participants) | 10
percentage of participants | 70

2. Secondary Outcome: Percentage of Participants With Decrease in 4E-binding protein1 (p4EBP1) Protein Phosphorylation From Baseline
Description: Percentage of men with downstream target inhibition of phosphatidylinositol 3-kinase (PI3K) in prostate tumor tissue as measured by 4E-binding protein1 (4EBP1) protein phosphorylation immunohistochemistry (IHC) using paired tumor biopsies from before and after drug administration and defined as >= 60% decline in p4EBP1 IHC
Time Frame: Up to 3 months
Population: One patient did not have pretreatment tissue evaluable for IHC
Measure: Number; unit: percentage of participants
Arm/Group | Neoadjuvant BKM120
Number analyzed (Participants) | 10
percentage of participants | 100

3. Secondary Outcome: Percentage of Participants With Decrease in AKT Protein From Baseline
Description: Proportion of men with downstream target inhibition of PI3K in prostate tumor tissue as measured by Protein kinase B (pAKT) IHC determined by a >= 60% decline in pAKT IHC
Time Frame: Up to 3 months
Population: One patient did not have pretreatment tissue evaluable for IHC
Measure: Number; unit: percentage of participants
Groups:
- Neoadjuvant BKM120: Twenty four men will receive 2 weeks of daily BKM120 prior to having radical prostatectomy
  BKM120: Two weeks after confirmatory biopsy, patients will begin taking 100 mg/day of BKM120. BKM120 will be given at this dose level orally once daily for 14 days prior to radical prostatectomy. Radical prostatectomy will be performed on the day of the last dose of BKM120 at day 14. No further drug will be administered after radical prostatectomy. For unforeseen delays in OR scheduling, up to 7 additional days of BKM120 may be administered prior to surgery.
Arm/Group | Neoadjuvant BKM120
Number analyzed (Participants) | 10
percentage of participants | 70

4. Secondary Outcome: Number of Participants Displaying Activity of Short Term BKM120 Administration
Description: Activity of short term BKM120 administration in prostate cancer was determined by measured PSA response immediately prior to radical prostatectomy
Time Frame: 1 Day, immediately prior to surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant BKM120
Number analyzed (Participants) | 11
Participants | 0

ADVERSE EVENTS:
Time Frame: Up to 3 months
Description: All adverse events, with severity/grading as determined by the NCI Common Terminology Criteria for Adverse Events (CTCAE).
Arm/Group | Neoadjuvant BKM120
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 3/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant BKM120 (N=11)
Irritability (General disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was closed early due to low accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes